CLINICAL TRIAL: NCT03022864
Title: Establishment of Accurate Diagnosis and Treatment System for Postoperative Chronic Pain Based on Functional Magnetic Resonance Imaging
Brief Title: Accurate Diagnosis System for Postoperative Chronic Pain Based on fMRI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MRI20161121
Record Dates: First submitted 2017-01-08; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Pain; Mammary Cancer
MeSH Terms: conditions — Chronic Pain; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic pain: Follow up the patients for three months after surgery using the designed table. If the patient evaluate the pain more than 3 points according the Numerical Rating Scale, then it can be considered that the patient has chronic pain.
- No chronic pain: Follow up the patients for three months after surgery using the designed table. If the patient evaluate the pain no more than 3 points according the Numerical Rating Scale, then it can be considered that the patient doesn't have chronic pain.

SUMMARY:
Postoperative pain is an ideal model for study on acute pain changing into chronic pain. The functional imaging of magnetic resonance can reflect the extent and character of pain exactly and the structural imaging of it can be a sign of the change. By analyzing fMRI results of participants with acute pain and following them up for three months, the investigators expect to find objective indicators for acute pain changing into chronic pain and give preventive analgesia for people with high risk of chronic pain.

DETAILED DESCRIPTION:
The day before surgery, evaluate and choose patients according to inclusion and exclusion criteria. Use the same anaesthesia and management and record information needed by the case report format. Patients are examined by fMRI on their brains during the first week after surgery. Follow up the patients after surgery for three months to find out whether they have chronic pain. The NRS, DN4, ID pain and QLQ-C30 are used for each patient.

ELIGIBILITY:
Inclusion Criteria:

* junior high school degree or above
* can be communicated in mandarin normally
* selective operation of mastectomy with or without axillary lymph node dissection
* similar operation method and incision size
* BMI between 18 and 30
* ASA grade I-II；informed consent

Exclusion Criteria:

* with brain disease or with brain disease history
* Opioid allergy
* with claustrophobia
* with history of chronic pain
* with psychological or emotional problems
* Serious hearing or visual impairment
* those who refuse to participant in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people who undergo selective operation of mastectomy with or without axillary lymph node dissection in ambulatory operation room of Shanghai RenJi Hospital （East part ) during year 2016 to 2018
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-11 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
different fMRI results of specific brain regions between people with and without chronic pain | in the first week after surgery
  amplitude of low frequency fluctuation(ALFF) and regional homogeneity(ReHo) of related brain regions

SECONDARY OUTCOMES:
the incidence of chronic pain after mastectomy | six months after surgery
  calculate the percentage of participants who rate pain more than three points on numerical rating scale
the quality of life in patients after mastectomy | six months after surgery
  the results of brief pain inventory in the first week after surgery and the EORTC QLQ-C30 results in the first, second and third month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Yu, Doctor, Study Chair — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apkarian AV, Bushnell MC, Treede RD, Zubieta JK. Human brain mechanisms of pain perception and regulation in health and disease. Eur J Pain. 2005 Aug;9(4):463-84. doi: 10.1016/j.ejpain.2004.11.001. Epub 2005 Jan 21. PMID 15979027
- [Background] Bailly F, Maigne JY, Genevay S, Marty M, Gandjbakhch F, Rozenberg S, Foltz V. Inflammatory pain pattern and pain with lumbar extension associated with Modic 1 changes on MRI: a prospective case-control study of 120 patients. Eur Spine J. 2014 Mar;23(3):493-7. doi: 10.1007/s00586-013-3036-6. Epub 2013 Sep 25. PMID 24221918
- [Background] Baliki MN, Geha PY, Fields HL, Apkarian AV. Predicting value of pain and analgesia: nucleus accumbens response to noxious stimuli changes in the presence of chronic pain. Neuron. 2010 Apr 15;66(1):149-60. doi: 10.1016/j.neuron.2010.03.002. PMID 20399736